CLINICAL TRIAL: NCT04321096
Title: The Impact of Camostat Mesilate on COVID-19 Infection: An Investigator-initiated Randomized, Placebo-controlled, Phase IIa Trial
Brief Title: The Impact of Camostat Mesilate on COVID-19 Infection
Acronym: CamoCO-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-001200-42
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Infection
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — camostat

STUDY DESIGN:
Intervention Model Description: There are 2 cohorts: Cohort 1 - hospitalized patients (n=180); Cohort 2 - outpatients (n=400). All participants in the two cohorts are randomized to one of two arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 2 pills 3 times daily for 5 days
  Interventions: Drug: Placebo oral tablet
- Camostat Mesilate (Experimental): 2x100 mg pills 3 times daily for 5 days
  Interventions: Drug: Camostat Mesilate

INTERVENTIONS:
Drug: Camostat Mesilate — Serine protease inhibitor that blocks TMPRSS-2 mediated cell entry of SARS-CoV-2
  Other Names: Foipan
  Arms: Camostat Mesilate
Drug: Placebo oral tablet — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
SARS-CoV-2, one of a family of human coronaviruses, was initially identified in December 2019 in Wuhan city. This new coronavirus causes a disease presentation which has now been named COVID-19. The virus has subsequently spread throughout the world and was declared a pandemic by the World Health Organisation on 11th March 2020. As of 18 March 2020, there are 198,193 number of confirmed cases with an estimated case-fatality of 3%. There is no approved therapy for COVID-19 and the current standard of care is supportive treatment.

SARS-CoV-2 exploits the cell entry receptor protein angiotensin converting enzyme II (ACE-2) to access and infect human cells. The interaction between ACE2 and the spike protein is not in the active site. This process requires the serine protease TMPRSS2. Camostat Mesilate is a potent serine protease inhibitor. Utilizing research on severe acute respiratory syndrome coronavirus (SARS-CoV) and the closely related SARS-CoV-2 cell entry mechanism, it has been demonstrated that SARS-CoV-2 cellular entry can be blocked by camostat mesilate. In mice, camostat mesilate dosed at concentrations similar to the clinically achievable concentration in humans reduced mortality following SARS-CoV infection from 100% to 30-35%.

DETAILED DESCRIPTION:
Cohort 1 - enrolment into the cohort of hospitalized patients has been completed (31 Dec 2020). Study results are publicly available at EClinicilMedicine, see link https://www.thelancet.com/journals/eclinm/article/PIIS2589-5370(21)00129-2/fulltext Cohort 2 - outpatients - remains open for enrolment

ELIGIBILITY:
Cohort 1)

* Documented COVID-19 infection as evidenced by positive PCR (or comparable clinical assay) for SARS-CoV-2
* Less than 48 hours since time of hospital admission OR if hospital-acquired COVID-19 is suspected, less than 48 hrs since onset of symptoms
* Adolescents and adults age >=18 years
* Subject or legally authorized representative able to give informed consent
* Admitted to hospital

Cohort 2)

* Documented COVID-19 infection as evidenced by positive PCR (or comparable clinical assay) for SARS-CoV-2
* One or more of the following symptoms of COVID-19 infection: fever, cough, expectoration, shortness of breath, myalgia, fatigue, or head ache
* No more than 5 days since the beginning of symptom onset
* Adolescents and adults age >=18 years
* Subject (or legally authorized representative, for Cohort 1 only) able to give informed consent
* Do not require immediate hospitalization (newly diagnosed COVID-19 patients who are discharged within 24 hrs of hospital admission are eligible for enrollment)
* Must be willing to fill out a daily symptom diary
* Must be available for a daily phone call
* Must be willing to take their own temperature at least once a day

Exclusion criteria

* Any condition that, in the Investigator's opinion, will prevent adequate compliance with study therapy (e.g. the patient is considered to be moribund within the next 72 hrs or has uncontrolled substance abuse that prevents adherence to study medication). Patients needing ventilator treatment are eligible to be enrolled if they fulfill the other in/exclusion criteria.
* The following laboratory values at baseline (Day 0):

  * Serum total bilirubin ≥3 ULN
  * Estimated glomerular filtration rate (eGFR) ≤30 mL/min (based on serum creatinine)
* Known hypersensitivity to Camostat Mesilate
* Women who are pregnant or breastfeeding, or with a positive pregnancy test as determined by a positive urine or blood beta- human chorionic gonadotropin test during screening or women of child bearing potential* who are unwilling or unable to use an acceptable method of contraception (combined estrogen and progestogen hormonal contraception (oral, intravaginal or transdermal), progesteron-only hormonal contraception (oral, injectable or implantable), intrauterine device or intrauterine hormone-releasing system) to avoid pregnancy during the study. Sexual abstinence will only be accepted in cases where this reflect the usual lifestyle.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Days to clinical improvement from study enrolment | 30 days
  Clinical improvement defined as live hospital discharge OR a 2 point improvement (from time of enrolment) in disease severity rating on the 7-point ordinal scale
Cohort 2: Days to clinical improvement from study enrolment | 30 days
  Days to clinical improvement from study enrolment defined no fever for at least 48 hrs AND improvement in other symptoms (e.g. cough, expectoration, myalgia, fatigue, or head ache)

SECONDARY OUTCOMES:
Safety evaluation, as measured by AEs, Adverse Reactions (ARs), SAEs, Serious ARs (SARs) | 30 days
Cohort 1: Clinical status as assessed by the 7-point ordinal scale at day 7, 14 and 30 | 30 days
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Cohort 1: Day 30 mortality | 30 days
  Mortality
Cohort 1: Change in NEW(2) score from baseline to day 30 | 30 days
  NEWS2
Cohort 1: Admission to ICU | 30 days
  ICU
Cohort 1: Use of invasive mechanical ventilation or ECMO | 30 days
  invasive mechanical ventilation or ECMO
Cohort 1: Duration of supplemental oxygen (days) | 30 days
  Nasal or high-flow oxygen
Cohort 1+2: Days to self-reported recovery (e.g. limitations in daily life activities) during telephone interviews conducted at day 30 | 30 days
  Subjective clinical improvement
Cohort 2: Number participant-reported secondary infection of housemates | 30 days
  No of new COVID-19 infections in the household
Cohort 2: Time to hospital admission related to COVID-19 infection | 30 days
  Hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Lars Østergaard, Professor, Study Chair — Head of Department
Locations (11):
- Denmark (10):
  - Region Hospital North Jutland, Hjørring, Region Nord
  - Department of Infectious Diseases, Aalborg
  - Department for Infectious Diseases, Aarhus University Hospital, Aarhus N
  - Bispebjerg hospital, Copenhagen
  - Herning Regional Hospital, Herning
  - Northzealands hospital - Hillerød, Hillerød
  - Horsens Regional Hospital, Horsens
  - Dept. of Infectious Diseases, Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Silkeborg Hospital, Silkeborg
- Örebro Hsopital, Örebro, Örebrolan, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan: Individual deidentified participant data (including data dictionaries) will be shared following the publication of the primary and secondary endpoints as outlined in this protocol. Data to be shared includes deidentified data points in published, peer-reviewed articles. Additional, related documents will also be available (study protocol, informed consent form, statistical analysis plan). Data will become available following publication with no planned end date.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Access to the data sharing will be given to researchers who provide a methodologically sound proposal for any type of analysis and requires IRB/Ethics committee approval (if applicable). Proposals should be addressed to olesoega@rm.dk.

REFERENCES:
- [Derived] Gunst JD, Staerke NB, Pahus MH, Kristensen LH, Bodilsen J, Lohse N, Dalgaard LS, Bronnum D, Frobert O, Honge B, Johansen IS, Monrad I, Erikstrup C, Rosendal R, Vilstrup E, Mariager T, Bove DG, Offersen R, Shakar S, Cajander S, Jorgensen NP, Sritharan SS, Breining P, Jespersen S, Mortensen KL, Jensen ML, Kolte L, Frattari GS, Larsen CS, Storgaard M, Nielsen LP, Tolstrup M, Saedder EA, Ostergaard LJ, Ngo HTT, Jensen MH, Hojen JF, Kjolby M, Sogaard OS. Efficacy of the TMPRSS2 inhibitor camostat mesilate in patients hospitalized with Covid-19-a double-blind randomized controlled trial. EClinicalMedicine. 2021 May;35:100849. doi: 10.1016/j.eclinm.2021.100849. Epub 2021 Apr 22. PMID 33903855